CLINICAL TRIAL: NCT00957463
Title: Effects of Intermittent Hypoxia and/or Cigarette Smoking on Endothelial Injury in Vivo - Relevance to Obstructive Sleep Apnea
Brief Title: Effects of Obstructive Sleep Apnea and/or Cigarette Smoking on Endothelial Function
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Mary SM Ip, The University of Hong Kong
Other Study IDs: UW 08-023
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Obstructive Sleep Apnea; Smoking
Keywords: endothelial function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- smoker, with high apnea-hypopnea index: subjects who smoke either in the past or currently, with confirmed moderate-severe OSA
- smoker, mild OSA or without OSA: subjects who smoke either in the past or currently, with mild OSA or without OSA
- nonsmoker, with high apnea-hypopnea index: subjects who never smoke, with confirmed moderate-severe OSA
- nonsmoker, with mild OSA or without OSA: subjects who never smoke, with mild OSA or without OSA

SUMMARY:
The hypothesis of this study is that either obstructive sleep apnea (OSA) or cigarette smoking (CS) exposure would produce oxidative stress and inflammation leading to endothelial injury, and the combined exposure would be additive or synergistic.

ELIGIBILITY:
Inclusion Criteria:

* No acute illness
* No hospitalization in past 4 weeks
* Absence of medical comorbidity such as hypertension, ischemic heart disease, diabetes and hyperlipidemia, renal impairment, vasculitis or Raynaud's syndrome, peripheral vascular disease especially Buerger's disease, aortic disease (aortic aneurysm or dilatation), cancer, thrombocytopenia, coagulation disorder or other chronic medical illness

Exclusion Criteria:

* Mentally incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects who undergo polysomnograms (PSG) in the Sleep Disorder Centre, Department of Medicine, Queen Mary Hospital, and who fulfill the study criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
reactive hyperemia induced peripheral arterial tone (RH-RAT) index | baseline

SECONDARY OUTCOMES:
circulatory metabolic and vascular inflammatory biomarkers | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mary SM Ip, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Barnoya J, Glantz SA. Cardiovascular effects of secondhand smoke: nearly as large as smoking. Circulation. 2005 May 24;111(20):2684-98. doi: 10.1161/CIRCULATIONAHA.104.492215. PMID 15911719
- [Background] Kashyap R, Hock LM, Bowman TJ. Higher prevalence of smoking in patients diagnosed as having obstructive sleep apnea. Sleep Breath. 2001 Dec;5(4):167-72. doi: 10.1007/s11325-001-0167-5. PMID 11868156
- [Background] Lavie L, Lavie P. Smoking interacts with sleep apnea to increase cardiovascular risk. Sleep Med. 2008 Mar;9(3):247-53. doi: 10.1016/j.sleep.2007.03.018. Epub 2007 May 21. PMID 17513169
- [Background] El Solh AA, Akinnusi ME, Baddoura FH, Mankowski CR. Endothelial cell apoptosis in obstructive sleep apnea: a link to endothelial dysfunction. Am J Respir Crit Care Med. 2007 Jun 1;175(11):1186-91. doi: 10.1164/rccm.200611-1598OC. Epub 2007 Feb 1. PMID 17272785
- [Background] Bernhard D, Wang XL. Smoking, oxidative stress and cardiovascular diseases--do anti-oxidative therapies fail? Curr Med Chem. 2007;14(16):1703-12. doi: 10.2174/092986707781058959. PMID 17627508
- [Background] Itzhaki S, Lavie L, Pillar G, Tal G, Lavie P. Endothelial dysfunction in obstructive sleep apnea measured by peripheral arterial tone response in the finger to reactive hyperemia. Sleep. 2005 May;28(5):594-600. doi: 10.1093/sleep/28.5.594. PMID 16171272